CLINICAL TRIAL: NCT04665921
Title: A Phase 1 Study of SGN-STNV in Advanced Solid Tumors
Brief Title: A Study of SGN-STNV in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGNSTNV-001
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Carcinoma, Non-Small Cell Lung; HER2 Negative Breast Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Gastroesophageal Junction Carcinoma; Stomach Neoplasms; Colorectal Neoplasms; Exocrine Pancreatic Adenocarcinoma; Appendiceal Adenocarcinoma; Pseudomyxoma Peritonei
Keywords: NSCLC; Non-Small Cell Lung Cancer; HER2-Negative Breast Cancer; High-Grade Serous Ovarian Cancer; HGSOC; Ovarian Cancer; Cervical Cancer; Endometrial Cancer; Esophageal Cancer; Gastric Cancer; GEJ Carcinoma; Colorectal Cancer; Seattle Genetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Adenocarcinoma, Mucinous; Pseudomyxoma Peritonei

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SGN-STNV (Experimental): SGN-STNV monotherapy
  Interventions: Drug: SGN-STNV

INTERVENTIONS:
Drug: SGN-STNV — Given into the vein (IV; intravenously)

SUMMARY:
This trial will look at a drug called SGN-STNV to find out whether it is safe for patients with solid tumors. It will study SGN-STNV to find out what its side effects are. A side effect is anything the drug does besides treating cancer. It will also study how well SGN-STNV works to treat solid tumors.

The study will have two parts. Part A of the study will find out how much SGN-STNV should be given to patients. Part B will use the dose found in Part A to find out how safe SGN-STNV is and if it works to treat certain types of solid tumors.

DETAILED DESCRIPTION:
The study will include dose escalation (Part A) and dose expansion (Part B), with multiple disease-specific cohorts and a biology cohort in dose expansion. The biology cohort will require additional biopsies. At the completion of dose escalation, up to 5 disease specific expansion cohorts and 1 biology expansion cohort may be activated by the sponsor in consultation with the Safety Monitoring Committee (SMC). Expansion cohorts in Part B will enroll subjects with selected tumors that are eligible for enrollment in Part A. The dose(s) to be examined in Part B will be at or below the maximum tolerated dose and/or the recommended dose determined in Part A. The recommended dose and/or schedule may differ between cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Disease indication

  * Must have disease that is relapsed or refractory or be intolerant to standard-of-care therapies and should have no appropriate standard-of-care therapeutic option.

    * Non-small cell lung cancer (NSCLC)
    * HER2 negative breast cancer
    * Ovarian cancer
    * Cervical cancer
    * Endometrial cancer
    * Esophageal cancer
    * Gastric cancer and GEJ carcinoma
    * Colorectal cancer
    * Exocrine pancreatic adenocarcinoma
    * Appendiceal adenocarcinoma and pseudomyxoma peritonei of unknown origin
* Participants enrolled in the following study parts should have an appropriate tumor site that satisfies the following criteria:

  * Site has tumor that is not a target lesion and has not been previously irradiated (unless progression has occurred since end of radiotherapy)
  * Site has tumor that is accessible for a minimally invasive biopsy that does not present a significant risk, AND
  * Participant must agree to a biopsy as follows

    * Disease-specific expansion cohorts: pre-treatment biopsy, unless medically infeasible following consultation with the medical monitor
    * Biology expansion cohort: pretreatment biopsy (required) and additional on-treatment biopsy during Cycle 1 (unless medically infeasible following consultation with the medical monitor)
* Measurable disease per the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) at baseline
* An Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Adequate renal, hepatic, and hematologic function

Exclusion Criteria

* History of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy.
* Known active central nervous system metastases
* Carcinomatous meningitis
* Previous receipt of monomethylauristatin E (MMAE)-containing drugs
* Pre-existing neuropathy ≥ Grade 2 per the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
* Any uncontrolled ≥ Grade 3 (per the NCI CTCAE, Version 5.0) viral, bacterial, or fungal infection within 2 weeks prior to the first dose of SGN-STNV

There are additional inclusion and exclusion criteria. The study center will determine if criteria for participation are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Through 30-37 days following last dose of SGN-STNV; up to approximately 3 years
  To be summarized using descriptive statistics
Incidence of laboratory abnormalities | Through 30-37 days following last dose of SGN-STNV; up to approximately 3 years
  To be summarized using descriptive statistics
Incidence of dose limiting toxicities | Up to 28 days
  To be summarized using descriptive statistics

SECONDARY OUTCOMES:
Objective response rate (ORR) as assessed by the investigator per RECIST v1.1 | Up to approximately 3 years
  ORR is defined as the proportion of subjects achieving a partial response (PR) or complete response (CR).
Progression-free survival (PFS) | Up to approximately 3 years
  PFS is defined as the time from the start of any study treatment to first documentation of disease progression or to death due to any cause, whichever comes first.
Overall survival (OS) | Up to approximately 3 years
  OS is defined as the time from the start of any study treatment to the date of death due to any cause.
Duration of objective response (DOR) | Up to approximately 3 years
  DOR is defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression or to death due to any cause, whichever comes first.
Area under the concentration-time curve (AUC) | Through 30-37 days following last dose of SGN-STNV; up to approximately 3 years
  Pharmacokinetic (PK) endpoint
Time to maximum concentration (Tmax) | Through 30-37 days following last dose of SGN-STNV; up to approximately 3 years
  PK endpoint
Maximum concentration (Cmax) | Through 30-37 days following last dose of SGN-STNV; up to approximately 3 years
  PK endpoint
Trough concentration (Ctrough) | Through 30-37 days following last dose of SGN-STNV; up to approximately 3 years
  PK endpoint
Incidence of antidrug antibodies (ADA) | Through 30-37 days following last dose of SGN-STNV; up to approximately 3 years
  Immunogenicity endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne McGoldrick, MD, Study Director — Seagen Inc.
Locations (18):
- United States (12):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of California, San Francisco | HDFCCC - Hematopoietic Malignancies, San Francisco, California
  - Shands Cancer Center / University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics Midwest, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- Canada (2):
  - University of Ottawa / Ottawa General Hospital, Ottawa, Ontario
  - University Health Network, Princess Margaret Hospital, Toronto, Other
- Institut Gustave Roussy, Villejuif, Other, France
- Istituto Europeo di Oncologia, Milan, Other, Italy
- Hospital Universitari Vall d'Hebron, Barcelona, Other, Spain
- The Royal Marsden Hospital (Surrey), Sutton, Other, United Kingdom